CLINICAL TRIAL: NCT07067619
Title: Pain Acceptance Training in Patients Experiencing Emotional Distress and Somatic Symptoms: Examination of Dialectical Thinking as a Mediating Factor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Rambam Hospital, Haifa, Israel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0062-24
Record Dates: First submitted 2025-07-01; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Somatic Pain; Comorbid Pain and Emotional Difficulties
Keywords: Chronic pain; Somatic pain; Pain Acceptance; Intervention; Training; Experimental pain
MeSH Terms: conditions — Chronic Pain; Nociceptive Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain-acceptance intervention group (Experimental): Patients in the pain-acceptance group will undergo a battery of baseline assessments in the first session, and receive a two-week intervention.
  First, they receive an explanation of pain acceptance, and practice it with the experimenter through discussion and metaphors, and do two exercises: STOP and a cold-pressor task.
  Next, they conduct two weeks of home practice. At home, they are asked to use the pain-acceptance strategy whenever they feel pain. After one week, the experimenter will conduct a short video call with the patient, to discuss the progress and the difficulties that arise in using the acceptance training.
  The experimenter also supports them by phone and video call as needed. Further, they complete a brief survey on pain, disability, strategy use, and ease on a daily base.
  After two weeks, they return for a follow-up assessment including questionnaires, cognitive tasks, and the cold-pressor test. Two weeks later they complete an online follow-up survey.
  Interventions: Behavioral: Pain-acceptance intervention
- treatment-as-usual group (No Intervention): Patients in the 'treatment as usual' will undergo a battery of baseline assessments in the first session, including questionnaires, cognitive task and Cold pressure task.
  Afterwards, they complete the daily online evaluations during two weeks. During this period, a brief online survey is sent to the participants daily in the evening via text massage. The survey include questions about pain severity and functional disability felt today. Additionally, at the end of the first week, they will have a video call with the experimenter , to discuses their feelings.
  At the end of the two-week pain evaluation, they will arrive for the end of intervention session of the assessments, and at the end of this session will be offered to receive the pain-acceptance intervention.
  Two weeks after the end of intervention assessment session, patients will receive a link to complete online the same battery of questionnaires as administered in the previous session.

INTERVENTIONS:
Behavioral: Pain-acceptance intervention — The intervention start with a conversation and inquiry about the participant's pain while continuously validating his experience and creating a shared understanding of their struggles and difficulties due to the pain.
  Next, the experimenter explain the relations between distress, pain and suffering, emphasizing that in many cases trying to control our pain, emotions and thoughts leads us to undesirable results through emotional avoidance, anger and escape. This explanation will be accompanied with commonly used metaphors to enhance participants' understanding. Afterwards, participants are familiarized with the strategy of "emotional acceptance of pain". The strategy will be comprehensively explained and participants will practice it with the experimenter twice: Firstly, by practicing with the mental exercise of "STOP" (i.e. Stop, Take a step back, Observe, Procced Mindfully); Secondly by practicing the pain acceptance strategy while feeling moderate pain, and discuss their experience.
  Arms: Pain-acceptance intervention group

SUMMARY:
Somatic symptoms, including physical pain, are highly prevalent among mental health patients. Current treatments have limited effectiveness for these symptoms, primarily because of patients' diminished introspective capacity and lack of emotional awareness. The current study proposes pain acceptance training as a new intervention. This intervention relies on the tenets of dialectical thinking, particularly on maintaining a dialectic perspective - at once acknowledging both the desire to end the pain and the ability to accept it as it is. We aim to examine the following: (1) the efficacy of pain acceptance training in the alleviation of somatic pain in patients with somatic symptoms; (2) the role of dialectical thinking as a mediator of pain acceptance training efficacy.

DETAILED DESCRIPTION:
Somatic symptom disorders are among the most common mental disorders, with an estimated prevalence of 5-7% in the general population1. Somatic disorders are characterized by persistent, unexplained physical symptoms, such as pain and gastrointestinal and cardiovascular symptoms, which cause significant impairments to regular functioning and high burden due to multiple medical consultations. A substantial proportion of patients also experience comorbid depression and anxiety.

Growing evidence indicates that specific maladaptive psychological factors (e.g., catastrophizing, emotion regulation problems, and negative physical self-concept) play a substantial role in causing and sustaining somatic symptoms. Therefore, psychological treatments such as cognitive behavioral therapy are the first line of treatment6. Still, individuals with somatic symptoms exhibit limited responsiveness to conventional psychotherapeutic approaches.

To remedy this, one possible approach is Dialectical Behavior Therapy (DBT), which aims to enhance dialectical thinking, a cognitive process that involves the ability to hold and reconcile opposing ideas or viewpoints and reflect on them curiously. Few studies have shown that increases in dialectical thinking during psychological treatment have positive effects on attention, coping flexibility, and self-processing.

A limited number of studies have examined the effects of DBT treatment among patients with somatic symptoms. One initial study exploring the effects of DBT in individuals suffering from somatic symptoms reported reduced somatization in patients diagnosed with borderline disorder, through an increase in emotional acceptance.

Though promising, DBT is a long-term, in-person intervention that must be carried out by trained professionals and is, therefore, resource-intensive and inaccessible to many people. Therefore, we propose an alternative related intervention for individuals experiencing somatic symptoms, namely Pain-Acceptance Training. Similar to DBT, the Pain-Acceptance Training targets core mechanisms related to pain processing and modulation.

CURRENT INTERVENTION

Pain-acceptance training is based on dialectical thinking, particularly in maintaining a dialectic perspective, on the suffering caused by the pain - simultaneously wishing it to end and accepting it. Acceptance-based pain interventions attempt to teach patients to experience their emotions, pains, and bodily sensations more fully and without avoidance, and to notice fully the presence of thoughts without following, resisting, believing, or disbelieving them. Accepting thoughts and feelings impedes the control these exert over behavioral tendencies and limits their impact on pursuing personal goals. Thus, even though acceptance-based strategies do not aim at pain reduction, various studies have shown that these strategies can alter the pain experience and therefore may be considered regulation strategies. This training method is also easily implemented, and can be imparted to participants both online and in person. Research shows that short trainings in pain acceptance regulation strategies increase pain tolerance, enhance recovery from pain, lower pain anxiety, distress ratings, and negative emotions related to pain, and facilitate better overall functioning despite the pain.

Prior Clinical Experience

In our recent randomized controlled single-session trial of pain-acceptance training that was conducted at the University of Haifa, healthy individuals showed reduced sensitivity to suprathreshold pain and reported an increase in pain threshold. This increase correlated with an increase in the vagal tone reactivity to pain, suggesting that the training modulates pain via the antinociceptive effect of the vagus nerve. Crucially and even more importantly, the reduction in pain sensitivity and increase in pain threshold were maintained for a month following the training, thus showing long long-lasting impact on pain perception. Furthermore, this training resulted in a decrease in pain catastrophizing levels one month later, suggesting that participants had better emotional capacities for dealing with pain.

RESEARCH OBJECTIVES & SIGNIFICANCE

As demonstrated, pain acceptance training showed promising results in altering the pain perception of healthy participants. The current study aims at translating these outcomes to a clinical setting; to examine a novel form of acceptance-training for pain relief in psychiatric patients suffering from somatic symptoms. We hypothesize that pain intensity, functional disability, and negative affect will decrease as a result of acceptance training, and that these changes will be mediated by an increase in patients' dialectical thinking abilities.

STUDY ENDPOINTS / OUTCOMES

To the best of our knowledge, this is the first study to examine pain acceptance training in psychiatric patients with somatic symptoms. To determine the efficacy of the training, we will utilize different pain outcome measures, and assess emotional and cognitive correlates of the change. As such, we believe this study will provide preliminary data that will serve as a basis for further randomized control trials examining the clinical implications of acceptance based training compared to other standard pain-treatment methods, and exploring the mechanisms underlying pain acceptance training for somatic symptoms relief.

Our primary training outcome measures will be pain-related, and will be conducted in three phases: Baseline, End of Intervention Assessments, and Follow-up Assessments. We expect that following two-week of acceptance training, patients will feel lower pain intensity and will show better abilities to cope with their pain. These improvements are expected to be maintained over time, and we will observe this in the follow up assessments.

These measures include pain intensity assessment, assessment of the degree of widespread body pain, pain catastrophizing levels and pain self-efficacy believes, as well as actual pain coping measurement of cold pain threshold, and cold pain tolerance.

The secondary training measures will include emotional state measures, dialectical thinking measures, and attention bias for pain. Demographic and medical records variables will serve as covariates for evaluating individual factors affecting training efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women
2. Aged 18-70
3. Able to provide a signed informed consent
4. Experiencing significant pain symptoms that interfere with daily-life functioning
5. Experiencing significant emotional distress symptoms

Exclusion Criteria:

Patients under the age of 18 and/or diagnosed with one or more of the following diagnoses will be excluded from participation in the study:

1. Patients rating their average pain in the last week and in the last month as less than 3 in a 0-10 numerical rating scale (i.e. NPS)
2. Patients rating their emotional distress levels as less than 25 in a 10-50 numerical rating scale (i.e. Kessler Psychological Distress Scale [K10])
3. Patients diagnosed with psychotic disorders and/or suffering from psychotic symptoms.
4. Patients diagnosed with Autism Spectrum disorder.
5. Patients diagnosed with Intellectual disability.
6. Patients diagnosed with eating disorders.
7. Patients with Immediate suicidal risk.
8. Patients who initiated a new drug and/or psychotherapy treatment within the last month.
9. Pregnant women.
10. Patients currently serving in the IDF.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Chronic pain levels | Measured at the baseline assessment session, at the evaluation session at the end of the two-weeks intervention, and after two weeks follow-up.
  Chronic pain levels will be measured by The BPI-SF is a validated and widely recommended tool for assessing pain severity and pain-related interference in chronic pain patients. It measures pain severity at its worst, least, average, and current level over the past week on a 0-10 scale, with 0 = no pain and 10 = worst pain imaginable. It also evaluates interference across seven domains (general activity, walking, work, mood, relations, sleep, and enjoyment of life), each scored 0-10, where 0 = no interference and 10 = complete interference. Scores can be averaged into the Pain Severity Index and Pain Interference Index. The BPI-SF is responsive to changes in pain over time.
Pain self-efficacy | Measured at the baseline assessment session, at the evaluation session at the end of the two-weeks intervention, and after two weeks follow-up.
  Measured by the Pain self-efficacy questionnaire (PSEQ). The PSEQ assesses the strength of a person's confidence in their ability to function, despite their pain. Patients are asked to rate how confident they are so that they can do each of the 10 activities or functions at present, despite their pain, by selecting a number on a seven-point scale, where zero equals 'not at all confident' and six equals 'completely confident'. Scores on the PSEQ may range from 0 to 60, with higher scores indicating stronger self-efficacy beliefs. Good reliability and validity of the PSEQ has been reported. The test-retest reliability and internal consistency of the PSEQ in two different studies with chronic pain patients were reported as 0.79 and 0.92, respectively.

SECONDARY OUTCOMES:
Depression levels | Measured at the baseline assessment session, at the evaluation session at the end of the two-weeks intervention, and after two weeks follow-up.
  Measured by using the Patient Health Questionnaire-9 (PHQ-9). A self-report questionnaire for adults, the purpose of which is to examine the presence and severity of clinical depression23. The questionnaire includes 9 items that are a list of major depressive symptoms, according to the DSM. For each item, the examinee is asked to estimate how often he was bothered by the statement described in the item during the last two weeks, on a 4-point Likert scale of 3 (0 - not at all, 3 - almost every day). In addition, the examinee was asked how much the problems he reported made it difficult for him to do his job, take care of things at home or get along with others. This last item is important and significant to assess the degree of distress caused to a person by his symptoms, and the score in it is closely related to the degree of the person's quality of life.
Anxiety levels | Measured at the baseline assessment session, at the evaluation session at the end of the two-weeks intervention, and after two weeks follow-up.
  Measured by using the Generalized Anxiety Disorder 7-Item Scale (GAD-7). A self-report questionnaire with 7 items describing anxiety symptoms. In this questionnaire, the participant is asked to describe how well each statement describes his situation in the past two weeks, on a 4-point Likert scale (0 - not at all, 3 - almost every day). The questionnaire is acceptable for use for research and clinical purposes to detect anxiety symptoms in general, and general anxiety symptoms in particular, both in the general population and in clinical populations. The questionnaire has good psychometric properties including high internal reliability (Cronbach's alpha index = 0.89), and high validity indices.
Dichotomous Thinking | Measured at the baseline assessment session, at the evaluation session at the end of the two-weeks intervention, and after two weeks follow-up.
  Measured by using the Dichotomous Thinking Inventory (DTI), a self-report measure used to assess a black-and-white cognitive thinking style or worldview. The questionnaire assesses an individual's dichotomous thinking style in a general setting by measuring the degree of positive view of dichotomy, such as dichotomous thinking being better than other thinking styles and dichotomy being consequent, deserved, and worthy. The DTI has 15 items scored on a 6-point scale ranging from 1 = disagree strongly to 6 = agree strongly. The DTI has 3 components: preference for dichotomy, dichotomous beliefs, and profit-and-loss thinking.
Daily pain ratings and pain disruption | Measured by evaluating daily pain ratings in the two weeks of the intervention period
  Measured by evaluating daily pain ratings in the two weeks during the intervention period, via online questionnaire, on a scale ranging from 0 -not pain at all, to 100 - maximum pain they can imagine. Further, evaluating who much the pain interfered with daily activities, on a scale ranging from 0 - not at all, to 100 - interfered with all daily tasks.
Perceived improvement following the intervention | Measured at the evaluation session at the end of the two-weeks intervention, and after two weeks follow-up.
  Measured by Patient's global impression of change (PGIC) scale. Patients rate their improvement on a seven-point scale, where 0 equals "very much worse" and 6 equals "very much improved". This scale will be asked only in the last session, at the end of the intervention period. Patients themselves make a subjective judgment about the meaning of the change to them following treatment, this scale is often taken as the external criterion or "gold standard" of clinically important change. However, this method, by itself, does not indicate what has improved.
Pain catastrophizing | Measured at the baseline assessment session, at the evaluation session at the end of the two-weeks intervention, and after two weeks follow-up.
  Measured by using the Pain catastrophizing scale (PCS). The PCS contains 13 items that measure catastrophic thoughts about pain in both clinical and non-clinical samples. Participants reflect on past painful experiences and indicate on a 5-point scale ranging from zero ("not at all") to four ("always") the degree to which they experience each of the 13 thoughts or feelings during the experience of a pain (i.e. "When I'm in pain it's terrible and I think it's never going to get any better"). Research has shown that the PCS is valid and reliable
Dialectical thinking | Measured at the baseline assessment session, at the evaluation session at the end of the two-weeks intervention, and after two weeks follow-up.
  Measured by the Dialectical Self Scale (DSS), a validated and reliable measure that assesses dialectical self-esteem as related to self-perception. The DSS is a 32-item instrument using a 7-point Likert scale ranging from strongly disagree to strongly agree to measure the perception of dialecticism. Sixteen items describe scenarios that are inconsistent with naive dialecticism which are reverse-scored to determine a dialectical self-esteem rating, with high scores representing greater degrees of dialecticism (i.e. individuals who are "more dialectically oriented").
Experimental pain threshold and tolerance | Measured at the baseline assessment session, and at the evaluation session at the end of the two-weeks intervention.
  Measured by using the Cold Pressor Task (CPT), which consists tub containing cold water. Water's temperature will be kept at 10-12°C, to create a moderate pain sensation. This is a usual temperature range when studying pain, and based on our vast experience with this task it appropriate for the present experiment. Participants will be seated in a chair adjacent to the container and asked to immerse their non-dominant hand into the tab for as long as they feel able to do so. Maximum duration of immersion will be five minutes.
  The outcome measure will be pain threshold, which indicates the number of seconds from immersion in the tub that the participant first reported feeling pain. Threshold is a behavioral index of hypervigilance towards the pain experienced in the cold pressure. The second outcome measure will be pain tolerance, which indicates the number of seconds from immersion in the tank that the participant can tolerate the pain
Attention bias to pain-related images | Measured at the baseline assessment session, at the evaluation session at the end of the two-weeks intervention, and after two weeks follow-up.
  Measured by the a computerized version of the emotional modification of the perceptual load paradigm. In this task, participants are required to indicate whether a target letter (X or N) appears on the screen, by responding to the corresponding letter on the keyboard.
  The task contains two perceptual load conditions, low and high, which are determined by the number of distracting letters appearing alongside the target letter. In the low load condition, one distracting letter appears on the screen alongside the target letter, whereas in the high load condition, four distracting letters appear on the screen together with the target letter. The distracting letters are chosen randomly from the letters K, H, V, Z, or W. The target and distracting letters appear randomly in six possible locations that create an imaginary circle at the center of the screen. The distracting pictures can be either neutral or pain-related one.
Daily anxiety, distress and mood | Measured by evaluating daily pain ratings in the two weeks of the intervention period
  Measured by evaluating daily anxiety, distress and mood ratings in the two weeks during the intervention period, via online questionnaires, asking how much the participants felt one of these feeling today on a scale ranging from 0 (not at all) to 100 (all the time).

OTHER OUTCOMES:
Usage and ease of usage in the pain-acceptance strategy | Measured by evaluating daily pain ratings in the two weeks of the intervention period
  Evaluating how much participants used the pain-acceptance strategy daily (ranging from 0 - never, to 100 - for all pain sensations), how easy was it for participants to use the strategy (ranging from 0 - not easy at all to use, to 100 - very easy to use), how much they perceive the strategy relief the pain (ranging from 0 - no relief at all, to 100 -maximum relief), and how much they perceive the strategy usage help them cope with the pain and the suffering (ranging from 0 - did not assist me coping with my pain, to 100 - assisted me greatly coping with my pain).

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Psychiatric Division, Rambam Health Care Campus, Haifa
  - University of Haifa, Haifa

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT07067619/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT07067619/ICF_001.pdf